CLINICAL TRIAL: NCT01634490
Title: Effects of Different Dietary Regimens on Tolerance Acquisition in Children With Cow's Milk Allergy
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Other Study IDs: 013908
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Cow's Milk Allergy
Keywords: cow's milk allergy; formulas; probiotics
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- infants receiving extensively hydrolysed casein formula: infants receiving extensively hydrolysed casein formula as substitutive formula
- extensively hydrolysed casein formula with Lactobacillus GG: infants receiving extensively hydrolysed casein with LGG as substitutive formula
- infants receiving rice hydrolyzed formula: infants receiving rice hydrolyzed formula as substitutive formula
- infants receiving soy-based formula: infants receiving soy-based formula as substitutive formula
- infants receiving amino-acid based formula: infants receiving amino-acid based formula as substitutive formula

SUMMARY:
Otherwise healthy infants (1-12 months of age at the diagnosis) with CMA were prospectively evaluated. Patients with cow's milk protein-induced anaphylaxis, eosinophilic disorders of the gastrointestinal tract, and food protein induced enterocolitic syndrome were excluded. A food challenge was performed 6 and 12 months after the diagnosis to assess clinical tolerance acquisition. Main demographic and clinical characteristics were collected for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy infants (1-12 months of age at the diagnosis) with cow's milk allergy were prospectively evaluated

Exclusion Criteria:

* Patients with cow's milk protein-induced anaphylaxis, eosinophilic disorders of the gastrointestinal tract, and food protein induced enterocolitic syndrome were excluded.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We prospectively evaluated otherwise healthy infants (1-12 months of age at the diagnosis) visit one the Pediatric Gastroenterology and Allergology Centre because of the necessity of a diagnostic oral food challenge for cow's milk proteins. Children were in stable clinical condition without signs of CMA already on exclusion diet with an hypoallergenic formula for a period of 7-15 days as presented by the general paediatrician, immediately the symptoms appear and before being attended at the Center for diagnosis of CMA.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the effect of different dietotherapeutic approaches on the time of tolerance acquisition in children with cow's milk allergy | about 4 year
  . Otherwise healthy infants (1-12 months of age at the diagnosis) with CMA were prospectively evaluated. Patients with cow's milk protein-induced anaphylaxis, eosinophilic disorders of the gastrointestinal tract, and food protein induced enterocolitic syndrome were excluded. A food challenge was performed 6 and 12 months after the diagnosis to assess clinical tolerance acquisition. Main demographic and clinical characteristics were collected for each patient.

REFERENCES:
- [Derived] Berni Canani R, Nocerino R, Terrin G, Frediani T, Lucarelli S, Cosenza L, Passariello A, Leone L, Granata V, Di Costanzo M, Pezzella V, Troncone R. Formula selection for management of children with cow's milk allergy influences the rate of acquisition of tolerance: a prospective multicenter study. J Pediatr. 2013 Sep;163(3):771-7.e1. doi: 10.1016/j.jpeds.2013.03.008. Epub 2013 Apr 10. PMID 23582142